CLINICAL TRIAL: NCT00712062
Title: Pilot Study to Determine Therapeutic Response of Pemetrexed (Alimta) in Recurrent or Progressive Primary Central Nervous System Lymphoma (PCNSL) by Establishing the Radiographic Response Rate Using Modified Macdonald Criteria
Brief Title: Study of Pemetrexed to Treat Recurrent or Progressive Primary Central Nervous System Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCNSL-001
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: PCNSL; Pemetrexed; Alimta; Recurrent; Progressive
MeSH Terms: conditions — Recurrence | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed (Experimental): 500 mg/m2 given as an injection into a vein over 10 minutes once every 21 days until progression or unacceptable toxicity.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 given as an injection into a vein over 10 minutes once every 21 days until progression or unacceptable toxicity.
  Other Names: Alimta

SUMMARY:
The purpose of this study is to determine if pemetrexed is effective in the treatment of primary central nervous system lymphoma (PCNSL) that has either worsened during treatment or has returned after completing treatment.

DETAILED DESCRIPTION:
Despite the aggressive upfront use of methotrexate-based chemotherapy, primary central nervous system lymphoma (PCNSL) almost uniformly results in recurrence or progression and death. Palliative chemotherapy offers an improvement in time-to-progression, symptom control, quality of life, and potentially, survival. However, no established chemotherapy regimen for recurrence exists and new treatments are needed. Pemetrexed is a rationale strategy for therapeutic palliation of recurrent or progressive PCNSL, given its mechanism of action, convenient administration, single agent efficacy, its well established management algorithms, and its evidence of safety and efficacy in systemic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of Primary Central Nervous System Lymphoma
* Male or female > 18 years of age or older
* Negative pregnancy test (if of childbearing potential)
* Any number of previous recurrences will be allowed
* Karnofsky Performance Status > 60
* Hematocrit > 30,000
* Platelet > 100,000
* Absolute Neutrophil Count > 1,500
* Bilirubin < 1.5 x upper limits of normal
* Transaminases (ALT and AST) < 1.5 x upper limits of normal
* Creatinine < 1.5 x upper limits of normal
* Creatinine Clearance > 45 mL/min
* Adequate medical health to participate in this study
* Adequate documentation of menopause (natural/surgical) or patient commitment to routine use of reliable birth control (barrier/hormonal)
* Ability to read and understand the patient informed consent form
* Ability and willingness to follow all requirements of the study including following all directions, taking medication as prescribed, and completion of all diaries and forms

Exclusion Criteria:

* Karnofsky Performance Status < 60
* Hematocrit < 30,000
* Platelet < 100,000
* Absolute Neutrophil Count < 1,500
* Bilirubin >1.5 x upper limits of normal
* Transaminases (ALT & AST) > 1.5 x upper limits of normal
* Creatinine > 1.5 x upper limits of normal
* Creatinine Clearance < 45 mL/min
* Inability to undergo gadolinium-contrasted MRIs, including severe claustrophobia or insufficient allergy prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Determine the therapeutic response of intravenous pemetrexed in recurrent or progressive primary central nervous system lymphoma by establishing the radiographic response rate using modified Macdonald criteria. | 2.5 Years

SECONDARY OUTCOMES:
Evaluate the longitudinal effect of intravenous pemetrexed on traditional quality of life and performance status measurements. | 2.5 Years
Evaluate the longitudinal tolerability of intravenous pemetrexed using standardized toxicity criteria. | 2.5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Dunbar, MD, Principal Investigator — University of Florida